CLINICAL TRIAL: NCT03615924
Title: A Randomised, Double-Blind, Parallel-Group, Multicentre, Phase III Study to Evaluate the Effect of Ticagrelor Versus Placebo in Reducing the Rate of Vaso-Occlusive Crises in Paediatric Patients With Sickle Cell Disease (HESTIA3)
Brief Title: Effect of Ticagrelor vs. Placebo in the Reduction of Vaso-occlusive Crises in Pediatric Patients With Sickle Cell Disease
Acronym: HESTIA3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recommendation from an independent data monitoring committee (DMC) and accepted by AstraZeneca.
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5136C00009
Record Dates: First submitted 2018-06-22; First posted 2018-08-06 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Sickle Cell Anemia; SCD; Platelet aggregation; Ticagrelor; Brilinta; VOC; Vaso-Occlusive Crises; ACS; painful crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor (Experimental): The double-blinded study drug dose will be weight dependent:
  * ≥12 to ≤24kg: Ticagrelor 15 mg, twice a day
  * >24 to ≤48 kg: Ticagrelor 30 mg, twice a day
  * >48 kg: Ticagrelor 45 mg, twice a day.
  Interventions: Drug: Ticagrelor
- Placebo (Placebo Comparator): The double-blinded study drug dose will be weight dependent:
  * ≥12 to ≤24kg: Placebo to match ticagrelor 15 mg, twice a day
  * >24 to ≤48 kg: Placebo to match ticagrelor 30 mg, twice a day
  * >48 kg: Placebo to match ticagrelor 45 mg, twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor — The double-blinded study drug dose will be weight dependent:
  * ≥12 to ≤24kg: Ticagrelor 15 mg, twice a day
  * >24 to ≤48 kg: Ticagrelor 30 mg, twice a day
  * >48 kg: Ticagrelor 45 mg, twice a day.
  Arms: Ticagrelor
Drug: Placebo — The double-blinded study drug dose will be weight dependent:
  * ≥12 to ≤24kg: Placebo to match ticagrelor 15 mg, twice a day
  * >24 to ≤48 kg: Placebo to match ticagrelor 30 mg, twice a day
  * >48 kg: Placebo to match ticagrelor 45 mg, twice a day.
  Arms: Placebo

SUMMARY:
The purpose of the study is to Evaluate the Effect of Ticagrelor versus Placebo in Reducing the Rate of Vaso-Occlusive Crises in Paediatric Patients with Sickle Cell Disease

DETAILED DESCRIPTION:
Hestia3 will evaluate the efficacy, safety and tolerability of ticagrelor versus placebo in children with SCD during treatment for at least 12 months and up to approximately 24 months.

* The target population are children aged ≥2 to <18 years of age and body weight of ≥12 kg diagnosed with HbSS or HbS/β0 confirmed by high-performance liquid chromatography or hemoglobin electrophoresis. At least 50 evaluable patients should be recruited in each of the age groups, ≥2 years to <12 years and ≥12 years to <18 years.
* To be eligible for the study, patients must have experienced at least 2 VOCs (defined as painful crisis and/or ACS) events in the past 12 months prior to Visit 1, indicating that the severity of the patient's disease justifies preventive chronic long-term treatment. The intent is to enroll only children aged 2 years or above, since VOCs become more frequent with age.
* Study participants should receive standard of care for SCD, adjusted to the individual patient at the discretion of the investigator, including routine health care screening examinations and immunizations according to local guidelines and health care programmers. Study drug will be given on the background of standard treatments for SCD. Study participants are not withheld from any other treatments that may be used in SCD (eg., hydroxyurea) during the trial, which is important considering the use of a placebo control group. However, restrictions apply to some medications and interventions that may be necessary for the patient's health and well-being during the study.
* Patients are to be followed up to 24 months or until a common study end date is reached defined as 12 months after the last patient is randomised. The expected average follow-up is 18 months. Considering inclusion of patients with at least 2 VOC events in the past year, this treatment duration is considered long enough to evaluate effects on VOC events as well as to capture safety and tolerability data supporting a potential future long term use of ticagrelor.
* Due to ticagrelor mechanism of action and the potential to reduce symptoms caused by ischemia during a vaso-occlusion, a composite endpoint with painful crises and/or ACS has been selected for the primary endpoint. Painful crisis is the most common reason for emergency department visits for patients with SCD with a significant impact on young patients' lives, affecting them physically and emotionally. Secondary endpoints are included to broaden the understanding of effects in patients with SCD and to also assess potential benefits on symptomatic disease burden and health-related quality of life (HRQL).
* Patients will be treated with 15, 30 and 45 mg bd or matching placebo, depending on body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent prior to any study specific procedures not part of standard medical care (local regulations and international guidelines are to be followed in determining the assent/consent requirements for children).
2. Male or female paediatric patients aged ≥2 to <18 years and body weight of ≥12 kg (at Visit 1), diagnosed with HbSS or HbS/β0 as confirmed by high-performance liquid chromatography or haemoglobin electrophoresis.

   Note: Diagnosis of SCD (if not confirmed prior to screening and records available on the medical file) should be confirmed for HbSS or HbS/β0 by high-performance liquid chromatography or haemoglobin electrophoresis, performed at the site's local lab, in order to confirm the type of mutation.
3. Have experienced at least 2 VOCs (painful crisis and/or ACS) as judged by the Investigator in the past 12 months prior to Visit 1. These VOCs need to be documented in the patient's medical records or in other documents that can be reconciled.
4. If ≤16 years old, must have had transcranial Doppler (TCD) within the past year prior to Visit 1. If this is not the case, a TCD examination must be done before proceeding in the study.
5. If ≥10 years old, must have had an ophthalmological examination within the past year prior to Visit 1. If this is not the case, the patient must be examined by an ophthalmologist before proceeding in the study. If local guidelines dictate ophthalmological examination at younger ages, those local guidelines should be followed.
6. If treated with hydroxyurea, the weight-adjusted dose must be stable for 3 months before screening.
7. Suitable venous access for the study-related blood sampling
8. Prior to dosing on day of randomisation (Visit 2), a negative urine (dipstick) pregnancy test performed at Screening (Visit 1) and at Visit 2 must be available for female patients of childbearing potential.
9. Females of childbearing potential (after menarche) must not become pregnant during study. Sexually active females must use a highly effective method of contraception which results in a low failure rate (ie, less than 1% per year). If use of effective contraception cannot be secured in sexually active females, the patient cannot be included in this study.

Exclusion Criteria:

1. History of transient ischaemic attack (TIA) or cerebrovascular accident (ischaemic or haemorrhagic), severe head trauma, intracranial haemorrhage, intracranial neoplasm, arteriovenous malformation, aneurysm, or proliferative retinopathy.
2. Findings on TCD: Current or previous values for time averaged mean of the maximum velocity (TAMMV) that are Conditional or Abnormal. Patients with Conditional TAMMV values or higher (≥153 cm/sec using TCD imaging technique [TCDi] which is corresponding to ≥170 cm/sec by the non-imaging technique). Both the middle cerebral artery and the internal carotid artery should be considered.

   Any other criteria that would locally be considered as TCD indications for chronic transfusion would also exclude the patient.
3. Active pathological bleeding or increased risk of bleeding complications according to Investigator
4. Haemoglobin <6 g/dL from test performed at Screening (Visit 1)
5. Platelets <100 x 10^9/L from test performed at Screening (Visit 1) Undergoing treatment with chronic red blood cell transfusion therapy.
6. Undergoing treatment with chronic red blood cell transfusion therapy.
7. Chronic use of NSAIDs defined as continuous intake >3 days per week that cannot be discontinued
8. Receiving chronic treatment with anticoagulants or antiplatelet drugs that cannot be discontinued
9. Moderate or severe hepatic impairment defined as laboratory values of alanine aminotransferase (ALT) >2 × upper limits of normal (ULN), total bilirubin >2 × ULN (unless judged by the Investigator to be caused by haemolysis), albumin <35 g/L (3.5 g/dL) and International normalised ratio (INR) >1.4, or symptoms of liver disease (eg, ascites) from test performed at Screening (Visit 1).
10. Renal failure requiring dialysis
11. Patient considered to be at risk of bradycardic events (eg, known sick sinus syndrome or second or third degree atrioventricular block) unless already treated with a permanent pacemaker.
12. Concomitant oral or intravenous therapy with strong or moderate cytochrome P450 3A (CYP3A) inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers, which cannot be stopped at least 5 half-lives before randomisation.
13. Active untreated malaria. Patients with suspected malaria at Screening (Visit 1) will be tested.
14. Known hypersensitivity or contraindication to ticagrelor
15. Patients who are currently pregnant or breastfeeding, or planning to become pregnant during the study or have given birth less than 3 months prior to Screening (Visit 1)
16. Any condition which, in the opinion of the Investigator, would make it unsafe or unsuitable for the patient to participate in this study
17. Concern for the inability of the patient or caregiver (defined as legally authorized representative) to comply with study procedures and/or follow-up
18. Previous randomisation in the present study.
19. Participation in another clinical study with an IP or device during the last 30 days preceding screening.
20. Involvement of member of patient's family, or patient self, in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 193 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Berggren, MD, PhD, Study Director — AstraZeneca; Matthew Heeney, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (48):
- United States (7):
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, Charleston, South Carolina
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Edegem
- Brazil (4):
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
- Egypt (4):
  - Research Site, Al Sharkeya
  - Research Site, Alexandria
  - Research Site, Cairo
  - Research Site, Dakahlia
- Ghana (3):
  - Research Site, Accra
  - Research Site, Ho
  - Research Site, Kumasi
- Research Site, Athens, Greece
- India (4):
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, Pune
  - Research Site, Wardha
- Italy (4):
  - Research Site, Catania
  - Research Site, Naples
  - Research Site, Padua
  - Research Site, Verona
- Kenya (3):
  - Research Site, Kisumu
  - Research Site, Nairobi
  - Research Site, Siaya
- Lebanon (2):
  - Research Site, Beirut
  - Research Site, Tripoli
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Soweto
- Spain (3):
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Madrid
- Research Site, Mbeya, Tanzania
- Turkey (Türkiye) (3):
  - Research Site, Antalya
  - Research Site, Mersin
  - Research Site, Seyhan
- Uganda (2):
  - Research Site, Kampala
  - Research Site, Masaka
- United Kingdom (3):
  - Research Site, Cardiff
  - Research Site, Glasgow
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Heeney MM, Abboud MR, Githanga J, Inusa BPD, Kanter J, Michelson AD, Nduba V, Musiime V, Apte M, Inati A, Taksande AM, Andersson M, Astrand M, Maklad N, Niazi M, Himmelmann A, Berggren AR. Ticagrelor vs placebo for the reduction of vaso-occlusive crises in pediatric sickle cell disease: the HESTIA3 study. Blood. 2022 Sep 29;140(13):1470-1481. doi: 10.1182/blood.2021014095. PMID 35849650
- [Derived] Heeney MM, Abboud MR, Amilon C, Andersson M, Githanga J, Inusa B, Kanter J, Leonsson-Zachrisson M, Michelson AD, Berggren AR; HESTIA3 study investigators. Ticagrelor versus placebo for the reduction of vaso-occlusive crises in pediatric sickle cell disease: Rationale and design of a randomized, double-blind, parallel-group, multicenter phase 3 study (HESTIA3). Contemp Clin Trials. 2019 Oct;85:105835. doi: 10.1016/j.cct.2019.105835. Epub 2019 Aug 22. PMID 31446143
- See also: Statistical Analysis Plan redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5136C00009&attachmentIdentifier=d032cbc0-d37d-4ecc-991e-c656722cee5a&fileName=D5136C00009(HESTIA)_Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=
- See also: Clinical Study Protocol redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5136C00009&attachmentIdentifier=1b352613-fe0a-427a-ab9f-b25f9922ac9c&fileName=D5136C00009(HESTIA)_Clinical_Study_Protocol_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III study was conducted in pediatric participants with sickle cell disease (SCD) at 53 sites in 16 countries (Kenya, India, Uganda, Egypt, Lebanon, Ghana, South Africa, Tanzania, United Kingdom, Turkey, Spain, Italy, Belgium, Greece, Brazil and United States) between 26 September 2018 and 13 August 2020.
Pre-assignment Details: Pediatric participants who experienced at least two vaso-occlusive crisis (VOC) events in the past 12 months prior to screening and who fulfilled the eligibility criteria were enrolled. Participants randomized to ticagrelor received doses based on weight band (at randomization): ≥12 to ≤24 kilogram (kg)=15 milligram (mg), >24 to ≤48 kg=30 mg, >48 kg=45 mg. A total of 193 participants were randomized in this study.
Groups:
- Ticagrelor 15/30/45 mg bd: Pediatric participants received ticagrelor 15 mg, or 30 mg, or 45 mg tablets orally twice daily (bd) for at least 12 months but no longer than 24 months. The dose of ticagrelor was determined based on body weight at randomization:
  * Participants with a body weight ≥12 to ≤24 kg received 1 tablet of ticagrelor 15 mg (1x15 mg) bd.
  * Participants with a body weight >24 to ≤48 kg received 2 tablets of ticagrelor 15 mg (2x15 mg) bd.
  * Participants with a body weight >48 kg received 3 tablets of ticagrelor 15 mg (3x15 mg) bd.
- Placebo: Pediatric participants received placebo matching with ticagrelor 15 mg, or 30 mg, or 45 mg tablets orally bd for at least 12 months but no longer than 24 months. The number of placebo tablets was determined based on body weight at randomization:
  * Participants with a body weight ≥12 to ≤24 kg received 1 tablet of placebo matching with ticagrelor 15 mg bd.
  * Participants with a body weight >24 to ≤48 kg received 2 tablets of placebo matching with ticagrelor 30 mg bd.
  * Participants with a body weight >48 kg received 3 tablets of placebo matching with ticagrelor 45 mg bd.
Period: Overall Study
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Started (Randomized to treatment.) | 101 | 92
Received Treatment | 101 | 92
Completed (Completed the study.) | 0 | 0
Not Completed | 101 | 92
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Randomized in error | 1 | 0
Not completed — Study termination by Sponsor | 94 | 86

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized participants regardless of treatment received.
Groups:
- Ticagrelor 15/30/45 mg bd: Pediatric participants received ticagrelor 15 mg, or 30 mg, or 45 mg tablets orally bd for at least 12 months but no longer than 24 months. The dose of ticagrelor was determined based on body weight at randomization:
  * Participants with a body weight ≥12 to ≤24 kg received 1 tablet of ticagrelor 15 mg (1x15 mg) bd.
  * Participants with a body weight >24 to ≤48 kg received 2 tablets of ticagrelor 15 mg (2x15 mg) bd.
  * Participants with a body weight >48 kg received 3 tablets of ticagrelor 15 mg (3x15 mg) bd.
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo | Total
Number analyzed (Participants) | 101 | 92 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.40 (4.128) | 10.12 (3.799) | 10.26 (3.967)
Age, Customized [Count of Participants; unit: Participants]
  ≥2 to <12 years | 61 | 54 | 115
  >=12 to <18 years | 40 | 38 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 43 | 91
  Male | 53 | 49 | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 21 | 46
  Black or African American | 60 | 51 | 111
  Asian | 15 | 15 | 30
  Other | 1 | 5 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 94 | 87 | 181

OUTCOME MEASURES:

1. Primary Outcome: Number of Vaso-Occlusive Crisis Events
Description: A VOC is the composite of a painful crisis and/or an acute chest syndrome (ACS) event. The number of VOC events is defined as the count of VOC events experienced by a participant throughout the treatment period.
Time Frame: From randomization (Day 0) up to end of study (EOS) visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: VOC events
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
VOC events | 249 | 202
Statistical Analysis 1: Comparison: Ticagrelor 15/30/45 mg bd vs Placebo; Incidence rates, incidence rate ratios, and p-values are from a negative binomial model analysis, with treatment group and baseline hydroxyurea use included in the model as covariates; Test type: Superiority; p = 0.7597, Negative binomial model; Incidence rate ratio = 1.06, 95% CI 2-sided [0.75 to 1.50]

2. Secondary Outcome: Number of Painful Crisis Events
Description: A painful crisis is an onset or worsening of pain that lasts at least 2 hours, for which there is no explanation other than vaso-occlusion and which requires therapy with oral or parenteral opioids, parenteral non-steroidal anti-inflammatory drugs, or other analgesics prescribed by a healthcare provider in a medical setting (such as a hospital, clinic or emergency room visit) or at home. Events with an onset date <=7 days of the previous event onset date are not counted as new events.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: painful crisis events
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
painful crisis events | 248 | 209
Statistical Analysis 1: Comparison: Ticagrelor 15/30/45 mg bd vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9037, Negative binomial model; Incidence rate ratio = 1.02, 95% CI 2-sided [0.72 to 1.45]

3. Secondary Outcome: Number of Acute Chest Syndrome Events
Description: The ACS is an acute illness characterized by fever and/or respiratory symptoms, accompanied by a new pulmonary infiltrate on a chest X-ray. Events with an onset date <=7 days of the previous event onset date are not counted as new events.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: ACS events
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
ACS events | 6 | 6
Statistical Analysis 1: Comparison: Ticagrelor 15/30/45 mg bd vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7136, Negative binomial model; Incidence rate ratio = 0.76, 95% CI 2-sided [0.17 to 3.30]

4. Secondary Outcome: Duration of Painful Crises
Description: The duration of painful crises is defined as the sum of the duration of painful crises experienced by a participant over the defined treatment period. If two or more events have overlapping durations, the overlapping days were counted only once.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: days
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
days | 1476 | 1441
Statistical Analysis 1: Comparison: Ticagrelor 15/30/45 mg bd vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4970, Negative binomial model; Incidence rate ratio = 0.84, 95% CI 2-sided [0.50 to 1.40]

5. Secondary Outcome: Number of Vaso-Occlusive Crisis Events Requiring Hospitalization or Emergency Department Visits
Description: The number of VOC events requiring hospitalization or emergency department visits is defined as the count of VOC events experienced by a participant over the treatment period, for which the primary setting for VOC treatment was in-patient hospitalization or emergency department. Events with an onset date <=7 days of the previous event onset date are not counted as new events.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: VOC events requiring hospitalization
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
VOC events requiring hospitalization | 87 | 51
Statistical Analysis 1: Comparison: Ticagrelor 15/30/45 mg bd vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1636, Negative binomial model; Incidence rate ratio = 1.43, 95% CI 2-sided [0.87 to 2.36]

6. Secondary Outcome: Number of Days Hospitalized for Vaso-Occlusive Crisis Events
Description: The number of days hospitalized for all individual VOC events experienced by a participant during the treatment period is defined as the sum of the duration of all individual hospitalizations (taking into account potential overlapping hospitalization days of VOC components) during VOC events experienced by a participant over the treatment period for which the primary setting for VOC treatment was in-patient hospitalization.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: days
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
days | 526 | 256
Statistical Analysis 1: Comparison: Ticagrelor 15/30/45 mg bd vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2011, Negative binomial model; Incidence rate ratio = 1.68, 95% CI 2-sided [0.76 to 3.75]

7. Secondary Outcome: Number of Acute Sickle Cell Disease Complications
Description: The number of acute SCD complications is defined as the count of all individual acute SCD complications experienced by a participant over the treatment period. Acute SCD complications are defined as any one or more of the following individual complications: Transient ischaemic attack/ischaemic stroke, hepatic sequestration, splenic sequestration, priapism, and dactylitis.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: acute SCD complications
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
acute SCD complications | 6 | 3

8. Secondary Outcome: Number of Days Hospitalized for Acute Sickle Cell Disease Complications
Description: The number of days hospitalized for acute SCD complications is defined as the sum of the duration of all individual hospitalizations (taking into account potential overlapping hospitalization days) due to acute SCD complications experienced by a participant over the treatment period, for which hospitalization was reported.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: days
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
days | 0 | 6
Statistical Analysis 1: Comparison: Ticagrelor 15/30/45 mg bd vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9940, Negative binomial model; Incidence rate ratio = 0.00, 95% CI 2-sided [lower limit 0.00] (Upper limit of confidence interval was not calculable due to 0 events in Ticagrelor 15/30/45 mg bd reporting group.)

9. Secondary Outcome: Number of Sickle Cell-Related Red Blood Cell (RBC) Transfusions
Description: The number of participants with at least one sickle cell-related RBC transfusion reported. Adverse events resulting in the need for RBC transfusions were captured prior to database lock to determine if the transfusion was sickle cell-related or not.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received.
Measure: Number; unit: RBC transfusions
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
RBC transfusions | 39 | 49
Statistical Analysis 1: Comparison: Ticagrelor 15/30/45 mg bd vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4822, Negative binomial model; Incidence rate ratio = 0.77, 95% CI 2-sided [0.38 to 1.58]

10. Secondary Outcome: Health-Related Quality of Life Total Score Using the Pediatric Quality of Life Inventory (PedsQL) Sickle Cell Disease Module
Description: The PedsQL SCD module instrument developed using a 5-point Likert scale (where 0= never and 4= almost always) for the participant self-report forms for ages ≥5 to <8 years, ≥8 to <13 years, and ≥13 to ≤18 years and the caregiver proxy-report form specific for ≥2 to <5 years was used. The PedsQL SCD module measures problems in the following categories:
  * Pain: 3 sub-scales
  * Worry: 2 sub-scales
  * Emotions: 1 sub-scale
  * Treatment: 1 sub-scale
  * Communication: 2 sub-scales
  * Total score PedsQL SCD module items were reverse-scored and linearly transformed to a 0 to 100 scale (0= 100, 1= 75, 2= 50, 3= 25, 4= 0) so that higher scores indicate better quality of life. To create the PedsQL SCD module total score (43/42/40 items - depending on version completed) the arithmetic mean of the transformed scores was computed as the sum of the items transformed scores divided by the number of items answered. Baseline values are the closest observation prior to and including the randomization visit.
Time Frame: For ages ≥2 to <5 years and ≥5 to <8 years: Baseline (observation prior to and including the randomization visit) and Months 6, and 12; For ages ≥8 to <13 years and ≥13 to ≤18 years: Baseline and Months 6, 12, and 18
Population: The FAS included all randomized participants regardless of treatment received. Only number of participants included in analysis at each time point are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
score on a scale
  >=2 to <5 years: Baseline: number analyzed (Participants) | 5 | 10
  >=2 to <5 years: Baseline | 88.81 (14.107) | 67.02 (20.041)
  >=2 to <5 years: Month 6: number analyzed (Participants) | 6 | 10
  >=2 to <5 years: Month 6 | 80.75 (20.779) | 81.37 (14.125)
  >=2 to <5 years: Month 12: number analyzed (Participants) | 0 | 1
  >=2 to <5 years: Month 12 |  | 88.10 (NA) — Standard deviation could not be calculated as only 1 participant had analyzable data.
  >=5 to <8 years: Baseline: number analyzed (Participants) | 24 | 14
  >=5 to <8 years: Baseline | 75.05 (20.147) | 74.04 (21.646)
  >=5 to <8 years: Month 6: number analyzed (Participants) | 23 | 14
  >=5 to <8 years: Month 6 | 83.04 (15.332) | 84.91 (18.117)
  >=5 to <8 years: Month 12: number analyzed (Participants) | 2 | 1
  >=5 to <8 years: Month 12 | 65.63 (48.614) | 97.50 (NA) — Standard deviation could not be calculated as only 1 participant had analyzable data.
  >=8 to <13 years: Baseline: number analyzed (Participants) | 31 | 46
  >=8 to <13 years: Baseline | 62.35 (24.725) | 67.98 (24.338)
  >=8 to <13 years: Month 6: number analyzed (Participants) | 28 | 43
  >=8 to <13 years: Month 6 | 76.52 (17.189) | 75.76 (21.749)
  >=8 to <13 years: Month 12: number analyzed (Participants) | 6 | 7
  >=8 to <13 years: Month 12 | 83.20 (13.479) | 64.12 (27.253)
  >=8 to <13 years: Month 18: number analyzed (Participants) | 1 | 0
  >=8 to <13 years: Month 18 | 86.05 (NA) — Standard deviation could not be calculated as only 1 participant had analyzable data. |
  >=13 to <=18 years: Baseline: number analyzed (Participants) | 37 | 22
  >=13 to <=18 years: Baseline | 64.45 (18.746) | 60.81 (24.979)
  >=13 to <=18 years: Month 6: number analyzed (Participants) | 36 | 20
  >=13 to <=18 years: Month 6 | 68.13 (16.811) | 74.42 (19.146)
  >=13 to <=18 years: Month 12: number analyzed (Participants) | 9 | 5
  >=13 to <=18 years: Month 12 | 63.05 (19.810) | 73.26 (22.589)
  >=13 to <=18 years: Month 18: number analyzed (Participants) | 1 | 0
  >=13 to <=18 years: Month 18 | 65.12 (NA) — Standard deviation could not be calculated as only 1 participant had analyzable data. |

11. Secondary Outcome: Fatigue Total Score Using Pediatric Quality of Life Inventory Multidimensional Fatigue Scale
Description: The PedsQL multidimensional fatigue scale instrument developed using a 5-point Likert scale (where 0= never and 4= almost always) for the participant self-report forms for ages ≥5 to <8 years, ≥8 to <13 years, and ≥13 to ≤18 years and the caregiver proxy-report form specific for ≥2 to <5 years was used. The PedsQL multidimensional fatigue scale measures problems in the following categories:
  * General (6 items)
  * Sleep/rest (6 items)
  * Cognitive fatigue (6 items)
  * Total score (18 items) PedsQL multidimensional fatigue scale items were reverse-scored and linearly transformed to a 0 to 100 scale (0= 100, 1= 75, 2= 50, 3= 25, 4= 0) so that higher scores indicate better quality of life. To create the PedsQL multidimensional fatigue scale total score (18 items), the arithmetic mean of the transformed scores was computed as the sum of the items transformed scores divided by the number of items answered. Baseline values are closest observation prior to and including randomization visit.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 101 | 92
score on a scale
  >=2 to <5 years: Baseline: number analyzed (Participants) | 5 | 10
  >=2 to <5 years: Baseline | 88.06 (16.304) | 70.56 (23.220)
  >=2 to <5 years: Month 6: number analyzed (Participants) | 5 | 10
  >=2 to <5 years: Month 6 | 84.44 (15.541) | 81.94 (22.775)
  >=2 to <5 years: Month 12: number analyzed (Participants) | 0 | 1
  >=2 to <5 years: Month 12 |  | 94.44 (NA) — Standard deviation could not be calculated as only 1 participant had analyzable data.
  >=5 to <8 years: Baseline: number analyzed (Participants) | 25 | 14
  >=5 to <8 years: Baseline | 82.33 (11.450) | 84.13 (16.139)
  >=5 to <8 years: Month 6: number analyzed (Participants) | 22 | 14
  >=5 to <8 years: Month 6 | 87.12 (10.553) | 87.70 (16.076)
  >=5 to <8 years: Month 12: number analyzed (Participants) | 2 | 1
  >=5 to <8 years: Month 12 | 95.83 (5.893) | 100.00 (NA) — Standard deviation could not be calculated as only 1 participant had analyzable data.
  >=8 to <13 years: Baseline: number analyzed (Participants) | 30 | 44
  >=8 to <13 years: Baseline | 64.72 (26.779) | 69.51 (25.261)
  >=8 to <13 years: Month 6: number analyzed (Participants) | 28 | 43
  >=8 to <13 years: Month 6 | 75.65 (18.571) | 77.89 (22.283)
  >=8 to <13 years: Month 12: number analyzed (Participants) | 6 | 7
  >=8 to <13 years: Month 12 | 81.48 (17.866) | 65.87 (25.495)
  >=8 to <13 years: Month 18: number analyzed (Participants) | 1 | 0
  >=8 to <13 years: Month 18 | 73.61 (NA) — Standard deviation could not be calculated as only 1 participant had analyzable data. |
  >=13 to <=18 years: Baseline: number analyzed (Participants) | 36 | 22
  >=13 to <=18 years: Baseline | 68.06 (21.781) | 67.17 (18.223)
  >=13 to <=18 years: Month 6: number analyzed (Participants) | 35 | 20
  >=13 to <=18 years: Month 6 | 73.53 (19.138) | 75.21 (14.913)
  >=13 to <=18 years: Month 12: number analyzed (Participants) | 9 | 5
  >=13 to <=18 years: Month 12 | 67.13 (22.556) | 60.28 (23.664)
  >=13 to <=18 years: Month 18: number analyzed (Participants) | 1 | 0
  >=13 to <=18 years: Month 18 | 72.22 (NA) — Standard deviation could not be calculated as only 1 participant had analyzable data. |

12. Secondary Outcome: Percentage of Days of Absence From School or Work Due to Sickle Cell Disease
Description: For participants attending school/work at randomization, absence from school/work due to SCD was recorded weekly by the participant in the eDevice with the help of the caregiver if needed. The percentage of days absent from school/work due to SCD in the defined treatment period was calculated as follows:
  Percentage of absent days = (total number of days reported)/(total number of questionnaires answered ×7).
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received. Only participants going to school or work at randomization are reported.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 94 | 82
percentage of days | 5.24 (8.942) | 4.24 (4.964)

13. Secondary Outcome: Average Intensity of Worst Pain Daily During Vaso-Occlusive Crisis Events in Participants <5 Years of Age
Description: The Face, Legs, Activity, Cry, Consolability (FLACC) scale is caregiver-reported and used to assess pain daily during the VOC event for those participants <5 years of age as determined at randomization. Each of the 5 behaviours observed are assigned a score of 0, 1 or 2. The total FLACC score ranges between 0 and 10, with 0 representing "no pain" and 10 representing "very much pain". Lower score indicate better outcome. Worst pain ratings were collected once daily throughout the duration of the VOC event using an eDevice.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received. Only participants <5 years of age who had experienced at least one individual VOC event and analyzed for pain assessment are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 3 | 5
score on a scale | 3.4 (2.51) | 2.9 (1.99)

14. Secondary Outcome: Average Intensity of Worst Pain Daily During Vaso-Occlusive Crisis Events in Participants ≥5 Years of Age
Description: The Faces Pain Scale-revised (FPS-R) was administered to assess pain daily during the VOC event by those participants aged ≥5 years as determined at randomization. The FPS-R consists of 6 faces and scoring ranges between 0 and 10 (with an increase in numeric value by 2), where 0 is "no pain" and 10 is "very much pain". Lower score indicate better outcome. Worst pain ratings were collected once daily throughout the duration of the VOC event using an eDevice.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received. Only participants ≥5 years of age who had experienced at least one individual VOC event and analyzed for pain assessment are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 44 | 40
score on a scale | 4.5 (2.71) | 4.1 (2.02)

15. Secondary Outcome: Type of Analgesics Used by Participants During Vaso-Occlusive Crisis Events
Description: Analgesics use (opioid and non-opioid) during VOC events.
Time Frame: From randomization (Day 0) up to EOS visit or date of premature study discontinuation, up to approximately 20 months
Population: The FAS included all randomized participants regardless of treatment received. Only participants who had at least one VOC and took an analgesic are reported.
Measure: Number; unit: participants
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 70 | 58
participants
  Opioids: Yes | 46 | 22
  Opioids: No | 57 | 50
  Non-opioids: Yes | 69 | 57
  Non-opioids: No | 14 | 7

16. Secondary Outcome: Palatability of the Study Treatment Assessed by Study Medication Palatability Assessment (SMPA) in Participants ≤4 Years of Age
Description: Response to palatability was assessed through the SMPA question "Was any behaviour observed when the study medication was given to this participant that would be indicative of a negative response to the palatability of the study medication?". This was presented as a binary outcome (that is, where "No" is no negative response and "Yes" is negative response). No negative response was considered as a positive outcome.
Time Frame: Baseline (randomization visit) and Month 6
Population: The Safety Analysis Set included all participants who received at least 1 single dose of randomized study treatment, ticagrelor or placebo, and for whom any post-dose data were available. Only participants ≤4 years of age who completed the assessment for study treatment palatability are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 6 | 10
Participants
  Baseline: Whole tablet: number analyzed (Participants) | 5 | 8
  Baseline: Whole tablet: Negative response to palatability - No | 5 | 8
  Baseline: Whole tablet: Negative response to palatability - Yes | 0 | 0
  Baseline: Dispersed tablet: number analyzed (Participants) | 1 | 2
  Baseline: Dispersed tablet: Negative response to palatability - No | 1 | 2
  Baseline: Dispersed tablet: Negative response to palatability - Yes | 0 | 0
  Month 6: Whole tablet: number analyzed (Participants) | 4 | 9
  Month 6: Whole tablet: Negative response to palatability - No | 4 | 9
  Month 6: Whole tablet: Negative response to palatability - Yes | 0 | 0
  Month 6: Dispersed tablet: number analyzed (Participants) | 1 | 1
  Month 6: Dispersed tablet: Negative response to palatability - No | 1 | 1
  Month 6: Dispersed tablet: Negative response to palatability - Yes | 0 | 0

17. Secondary Outcome: Swallowability of the Study Treatment Assessed by Study Medication Palatability Assessment in Participants ≤4 Years of Age
Description: An observer's assessment of the participant's behaviour using the SMPA was performed for all participants taking the study treatment who are 2 to 4 years of age. Willingness to swallow was assessed and categorized as follows:
  * Swallowed without a problem
  * Some resistance but did swallow
  * Spit out some/all of the medication
  * Vomited up the medication. The category "swallowed without a problem" was considered as positive outcome.
Time Frame: Baseline (randomization visit) and Month 6
Population: The Safety Analysis Set included all participants who received at least 1 single dose of randomized study treatment, ticagrelor or placebo, and for whom any post-dose data were available. Only participants ≤4 years of age who completed the assessment for study treatment swallowability are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 6 | 10
Participants
  Baseline: Whole tablet: number analyzed (Participants) | 5 | 8
  Baseline: Whole tablet: Swallow without problem | 5 | 8
  Baseline: Whole tablet: Some resistance but did swallow | 0 | 0
  Baseline: Whole tablet: Spit out some/all medication | 0 | 0
  Baseline: Whole tablet: Vomited up medication | 0 | 0
  Baseline: Dispersed tablet: number analyzed (Participants) | 1 | 2
  Baseline: Dispersed tablet: Swallow without problem | 1 | 2
  Baseline: Dispersed tablet: Some resistance but did swallow | 0 | 0
  Baseline: Dispersed tablet: Spit out some/all medication | 0 | 0
  Baseline: Dispersed tablet: Vomited up medication | 0 | 0
  Month 6: Whole tablet: number analyzed (Participants) | 4 | 9
  Month 6: Whole tablet: Swallow without problem | 4 | 9
  Month 6: Whole tablet: Some resistance but did swallow | 0 | 0
  Month 6: Whole tablet: Spit out some/all medication | 0 | 0
  Month 6: Whole tablet: Vomited up medication | 0 | 0
  Month 6: Dispersed tablet: number analyzed (Participants) | 1 | 1
  Month 6: Dispersed tablet: Swallow without problem | 1 | 1
  Month 6: Dispersed tablet: Some resistance but did swallow | 0 | 0
  Month 6: Dispersed tablet: Spit out some/all medication | 0 | 0
  Month 6: Dispersed tablet: Vomited up medication | 0 | 0

18. Secondary Outcome: Palatability of the Study Treatment Assessed by Facial Hedonic Scale (FHS) in Participants ≥5 Years of Age
Description: The FHS method was used for all participants taking the study treatment who are ≥5 years of age. The FHS consists of 5 faces with descriptions ranging from "Dislike very much" to "Like very much". The face with description "Like very much" was considered as positive outcome. The way in which the study treatment was taken, that is, whether the tablet is whole or dispersed, was captured.
Time Frame: Baseline (randomization visit) and Month 6
Population: The Safety Analysis Set included all participants who received at least 1 single dose of randomized study treatment, ticagrelor or placebo, and for whom any post-dose data were available. Only participants ≥5 years of age who completed the assessment for study treatment palatability are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
Number analyzed (Participants) | 93 | 82
Participants
  Baseline: Whole tablet: number analyzed (Participants) | 92 | 80
  Baseline: Whole tablet: Dislike very much | 3 | 2
  Baseline: Whole tablet: Dislike a little | 4 | 2
  Baseline: Whole tablet: Not sure | 12 | 8
  Baseline: Whole tablet: Like a little | 25 | 23
  Baseline: Whole tablet: Like very much | 48 | 45
  Baseline: Dispersed tablet: number analyzed (Participants) | 1 | 2
  Baseline: Dispersed tablet: Dislike very much | 0 | 0
  Baseline: Dispersed tablet: Dislike a little | 0 | 0
  Baseline: Dispersed tablet: Not sure | 1 | 0
  Baseline: Dispersed tablet: Like a little | 0 | 1
  Baseline: Dispersed tablet: Like very much | 0 | 1
  Month 6: Whole tablet: number analyzed (Participants) | 83 | 74
  Month 6: Whole tablet: Dislike very much | 0 | 0
  Month 6: Whole tablet: Dislike a little | 5 | 3
  Month 6: Whole tablet: Not sure | 4 | 4
  Month 6: Whole tablet: Like a little | 30 | 20
  Month 6: Whole tablet: Like very much | 44 | 47
  Month 6: Dispersed tablet: number analyzed (Participants) | 1 | 0
  Month 6: Dispersed tablet: Dislike very much | 0 |
  Month 6: Dispersed tablet: Dislike a little | 0 |
  Month 6: Dispersed tablet: Not sure | 1 |
  Month 6: Dispersed tablet: Like a little | 0 |
  Month 6: Dispersed tablet: Like very much | 0 |

ADVERSE EVENTS:
Time Frame: From first dose of study treatment (Day 0) up to 7 days after last dose of study treatment, approximately 20 months.
Description: The Safety Analysis Set included all participants who received at least 1 single dose of randomized study treatment, ticagrelor or placebo, and for whom any post-dose data were available.
Arm/Group | Ticagrelor 15/30/45 mg bd | Placebo
All-Cause Mortality (participants affected / at risk) | 3/100 | 1/92
Serious Adverse Events (participants affected / at risk) | 44/100 | 29/92
Other Adverse Events (participants affected / at risk) | 82/100 | 71/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 15/30/45 mg bd (N=100) | Placebo (N=92)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 7 (13)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 39 (75) | 24 (41)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (4)
Sudden death (General disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (3)
Malaria (Infections and infestations) | 4 (4) | 1 (2)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 15/30/45 mg bd (N=100) | Placebo (N=92)
Leukocytosis (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 60 (190) | 49 (176)
Abdominal pain (Gastrointestinal disorders) | 15 (35) | 10 (16)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 5 (5)
Vomiting (Gastrointestinal disorders) | 6 (8) | 2 (2)
Non-cardiac chest pain (General disorders) | 7 (10) | 5 (5)
Pain (General disorders) | 5 (18) | 8 (9)
Pyrexia (General disorders) | 11 (15) | 10 (12)
Gastroenteritis (Infections and infestations) | 6 (7) | 4 (5)
Malaria (Infections and infestations) | 12 (15) | 7 (8)
Nasopharyngitis (Infections and infestations) | 4 (7) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 19 (28) | 24 (33)
Urinary tract infection (Infections and infestations) | 2 (3) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (17) | 14 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (28) | 12 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (58) | 23 (39)
Headache (Nervous system disorders) | 24 (44) | 18 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 7 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 8 (13)

LIMITATIONS AND CAVEATS:
AstraZeneca took the decision to terminate the study early, following a recommendation from the independent Data Monitoring Committee. This early termination was not considered to have had an impact on the robustness of the study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT03615924/Prot_001.pdf
  • Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT03615924/SAP_002.pdf